CLINICAL TRIAL: NCT00953043
Title: The Effect of Lubiprostone, a Chloride Channel Activator, on Colonic Sensorimotor Functions in Healthy Subjects. A Phase IV, Placebo-Controlled, Parallel Group Study
Brief Title: Lubiprostone, Colonic Motility and Sensation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH); Takeda (Industry)
Responsible Party: Michael Camilleri, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-001438; K24DK002638 (NIH); R01DK054681 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2012-02-09 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: lubiprostone; colon; motility; sensation
MeSH Terms: interventions — Lubiprostone; Cathartics; polyethylene glycol 3350

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lubiprostone (Active Comparator): Subjects randomized to this arm received 24 micrograms of lubiprostone per day for three days.
  Interventions: Drug: lubiprostone; Other: Bowel preparation
- Placebo (Placebo Comparator): Subjects randomized to this arm received placebo medication for three days.
  Interventions: Drug: Placebo; Other: Bowel preparation

INTERVENTIONS:
Drug: lubiprostone — Lubiprostone 24 micrograms, one dose daily for three days in 30 subjects
  Other Names: Amitiza
  Arms: Lubiprostone
Drug: Placebo — Placebo medication given for three days
  Arms: Placebo
Other: Bowel preparation — Polyethylene glycol-based bowel preparation
  Other Names: NuLytely

SUMMARY:
This study is being done to evaluate the effects of lubiprostone, a drug approved and used for constipation, on pattern of contractions of the colon and the colon's sensitivity to distension.

DETAILED DESCRIPTION:
This was a trial of healthy adults to compare the effects of oral lubiprostone, 24 microgram per day and placebo for three days, on sensation and contractions of the colon using validated methods.

On days 1 and 2, participants took the study medication with their breakfast and recorded the time. On day 2 starting at 4:00 pm, participants started a polyethylene glycol-based bowel preparation to cleanse the colon. After overnight bowl preparation, participants reported fasting to the study center at 7:00 am on day 3. Colonic sensorimotor functions were assessed by an endoscopically placed barostat-manometric assembly.

After 30 minutes of rest following tube placement, fasting colonic tone, colonic compliance and colonic sensation were tested. The last dose of medication was ingested and 1 hour later the same colonic functions, as well as colonic response to a standardized meal of a 1,000-kilocalorie chocolate milkshake were assessed. The participant was able to leave the study center in the afternoon, after a meal had been ingested (if desired).

Details on colonic tube placement: A flexible sigmoidoscopy was performed to evaluate the left side of the colon and to place a Teflon-coated guide wire beyond the splenic flexure. The colon was deflated as the sigmoidoscope was removed and a barostat catheter (constructed at Mayo Clinic, Rochester, MN) with six manometric point sensors and a polyethylene balloon was introduced into the colon over the guide wire. The barostat catheter was positioned in the mid-descending or upper sigmoid colon with the aid of fluoroscopy. The final position of the barostatically controlled balloon was confirmed by fluoroscopy. After the colonic tube placement, participants rested for 30 min. The catheter was connected to a rigid piston barostat machine. After transient inflation of the barostat bag to a volume of 75 ml to ensure it was unfolded, it was deflated. Thereafter, it was inflated in 2 mm Hg increments to baseline operating pressure, which was defined as 2 mm Hg above the minimal distension pressure at which respiratory excursions were clearly recorded by the barostat tracing.

ELIGIBILITY:
Inclusion criteria:

* Healthy subjects
* Body mass index (BMI): 18 to 32.
* Negative pregnancy test for women of childbearing potential.
* Absence of gastrointestinal symptoms (abridged Bowel Disease Questionnaire).
* Signed informed consent.

Exclusion criteria:

* Subjects with body mass index (BMI) of less than 18 or more than 32.
* Structural or metabolic diseases/conditions that affect the gastrointestinal (GI)system, or functional gastrointestinal disorders. For screening, the Bowel Disease Questionnaire will be used to exclude subjects with irritable bowel syndrome.
* Use of drugs or agents within the past 2 weeks that alter GI transit including laxatives, magnesium or aluminum-containing antacids, prokinetics, erythromycin, narcotics, anticholinergics, tricyclic antidepressants, SSRI and newer antidepressants.

NOTE: Low stable doses of thyroid replacement, estrogen replacement, low dose aspirin for cardioprotection, and birth control pills or depot injections are permissible.

* Use of drugs or agents within the 2 weeks prior to screening that may add drowsiness and central nervous system (CNS) depression such as barbiturates, benzodiazepines, ethanol, lithium, opioids, buspirone, antihistamines, muscle relaxants, other CNS depressants.
* Female subjects who are pregnant or breast feeding.
* Females must be either surgically sterilized, postmenopausal (>12 months since last menses) or, if of childbearing potential, using reliable methods of contraception as determined by the physician (single-barrier methods alone and rhythm methods are not acceptable).
* Clinical evidence (including physical exam and ECG) of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric, or other disease that interfere with the objectives of the study. Any candidate participants with such disorder mentioned will be referred to their general physician.
* The Hospital Anxiety and Depression Scale (HADS) will be used to exclude subjects with significant affective disorders, as well as to determine anxiety and depression scores at the start of the study. Any candidate participants with such disorder mentioned will be referred to their general physician.
* Symptoms of a significant clinical illness in the two weeks prior to screening.
* Participation in another clinical study within the 30 days prior to screening.
* Subjects who are considered by the investigator to be alcoholics not in remission or known substance abusers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Sweetser S, Busciglio IA, Camilleri M, Bharucha AE, Szarka LA, Papathanasopoulos A, Burton DD, Eckert DJ, Zinsmeister AR. Effect of a chloride channel activator, lubiprostone, on colonic sensory and motor functions in healthy subjects. Am J Physiol Gastrointest Liver Physiol. 2009 Feb;296(2):G295-301. doi: 10.1152/ajpgi.90558.2008. Epub 2008 Nov 25. PMID 19033530

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between September 2007 and July 2008 at the Mayo Clinic, Rochester, Minnesota.
Period: Overall Study
Arm/Group | Lubiprostone | Placebo
Started | 30 | 30
Completed | 26 | 28
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lubiprostone | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age Continuous [Mean (Standard Deviation); unit: years] | 35.1 (2.31) | 33.2 (2.18) | 34.1 (1.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body mass index is defined as the individual's body weight divided by the square of his or her height.
  kg/m^2 | 25.3 (0.54) | 25.5 (0.74) | 25.4 (0.45)

OUTCOME MEASURES:

1. Primary Outcome: Colonic Compliance
Description: Colonic compliance is a measure of the "stiffness" of the colon, that is, what pressure was needed to reach half the maximum volume of the colon.
  After the barostat catheter was inserted in the colon, the catheter was connected to a barostat machine. After an initial conditioning distension to 20 mm Hg, colonic compliance was measured by step-wise inflation with increments of 4 mm Hg up to 64 mm Hg. Colonic compliance was analyzed by a validated linear interpolation method. The pressure at half maximum volume serves as a summary of colonic compliance.
Time Frame: 1 hour after third dose of lubiprostone or placebo, on Day 3
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 26 | 28
mm Hg | 16.60 (0.817) | 16.50 (0.842)

2. Primary Outcome: Fasting Colonic Tone
Description: Colonic tone is a measurement of the volume of the colon. Colonic tone was assessed by noting the changes in the balloon volume in the presence of a constant operating pressure in the balloon (in the barostat-manometric assembly placed in the colon).
Time Frame: 30 minutes after the colonic tube placement, on Day 3
Measure: Mean (Standard Error); unit: mL
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 26 | 28
mL | 101.9 (7.479) | 112.8 (6.068)

3. Primary Outcome: Postprandial Colonic Tone
Description: Colonic tone was assessed by noting the changes in the balloon volume in the presence of a constant operating pressure in the balloon (in the barostat-manometric assembly placed in the colon).
Time Frame: 30 minutes after standard meal, on Day 3
Measure: Mean (Standard Error); unit: mL
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 26 | 28
mL | 78.69 (6.202) | 75.01 (3.492)

4. Primary Outcome: Pain Sensation Ratings in Response to Colonic Distension at 32 mm HG Above Baseline Operating Pressure
Description: Pain was measured by a 100 mm long Visual Analog Scale (VAS). The VAS does not have any pre-set marks between the extremes of 0 for no pain and 100 mm for extreme pain. The investigator measures the mark made by the participant in mm and records this for the value of pain.
Time Frame: approximately 1 hour after colonic tube placement, on Day 3
Measure: Mean (Standard Error); unit: mm
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 26 | 28
mm | 55.2 (4.38) | 55.8 (4.16)

5. Secondary Outcome: Gas Sensation Ratings in Response to Colonic Distensions at 32 mm Hg Above Baseline Operating Pressure
Description: Gas sensation was measured by a 100 mm long Visual Analog Scale (VAS). The VAS does not have any pre-set marks between the extremes of 0 for no gas sensation and 100 mm for extreme gas sensation. The investigator measures the mark made by the participant in mm and records this for the value of gas sensation.
Time Frame: approximately 1 hour after colonic tube placement, on Day 3
Measure: Mean (Standard Error); unit: mm
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 26 | 28
mm | 51.4 (4.37) | 54.6 (4.48)

6. Secondary Outcome: Median Pressure When First Sensation Was Reported by 50% of Participants
Description: The sensory threshold for first sensation was measured by stepwise inflation in increments of 4 mm Hg at 60 second intervals up to a maximum pressure of 64 mmg Hg. During this assessment participants were asked to report when they had the first sensation. The investigator recorded the threshold pressure at which the participants reported this sensation.
Time Frame: approximately 45 min after colonic tube placement, on Day 3
Measure: Median (Full Range); unit: mm Hg
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 26 | 28
mm Hg | 16 [0 to 64] | 12 [0 to 64]

7. Secondary Outcome: Median Pressure When Gas Sensation Was First Reported by 50% of Participants
Description: The sensory threshold for first perception of gas was measured by stepwise inflation in increments of 4 mm Hg at 60 second intervals up to a maximum pressure of 64 mmg Hg. During this assessment participants were asked to report when they had the first perception of gas. The investigator recorded the threshold pressure at which the participants reported this sensation.
Time Frame: approximately 45 min after colonic tube placement, on Day 3
Measure: Median (Full Range); unit: mm Hg
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 26 | 28
mm Hg | 28 [0 to 64] | 24 [0 to 64]

8. Secondary Outcome: Median Pressure When Pain Sensation Was First Reported by 50% of Participants
Description: The sensory threshold for first perception of pain was measured by stepwise inflation in increments of 4 mm Hg at 60 second intervals up to a maximum pressure of 64 mmg Hg. During this assessment participants were asked to report when they had the first perception of pain. The investigator recorded the threshold pressure at which the participants reported this sensation.
Time Frame: approximately 45 min after colonic tube placement, on Day 3
Measure: Median (Full Range); unit: mm Hg
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 26 | 28
mm Hg | 44 [0 to 64] | 40 [0 to 64]

ADVERSE EVENTS:
Time Frame: 72 hours after completion of the study
Arm/Group | Lubiprostone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/28
Other Adverse Events (participants affected / at risk) | 1/26 | 2/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lubiprostone (N=26) | Placebo (N=28)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Light-headed (Nervous system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was conducted in healthy subjects and needs replication in patients with Irritable Bowel Syndrome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No